CLINICAL TRIAL: NCT02059018
Title: The Underlying Mechanisms of Diameter Changes in Retinal Vessels During Hypoxia
Brief Title: The Mechanisms of Diameter Changes in Retinal Vessels During Hypoxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HypNOCOX-2; 1-10-72-14-14 (Other: Local ethical committe for medical science)
Record Dates: First submitted 2014-02-07; First posted 2014-02-11 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2014-01

CONDITIONS: Retinal Hypoxia
MeSH Terms: interventions — Cyclooxygenase Inhibitors; Nitroglycerin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypoxia (Experimental): Inhaling hypoxic gas mixture to induce hypoxemia during recordings of diameter changes of retinal vessels. Recording are performed during hypoxia alone and in combination with the associated interventions over two examination days
  Interventions: Drug: COX-inhibitor; Drug: Nitroglycerin; Drug: COX-inhibitor + Nitroglycerin
- Normoxia (Experimental): Breathing atmospheric air during recordings of diameter changes of retinal vessels. Recording are performed during normoxia alone and in combination with the associated interventions over two examination days
  Interventions: Drug: COX-inhibitor; Drug: Nitroglycerin; Drug: COX-inhibitor + Nitroglycerin

INTERVENTIONS:
Drug: COX-inhibitor — Administration of 1 drop voltaren 45 minutes before recordings of diameter changes of retinal vessels are initiated
  Other Names: Eye drops diclofenac 1mg/ml; Voltaren eye drops
Drug: Nitroglycerin — Oral administration of tablet nitroglycerin 0,5mg 5 minutes before recordings of diameter changes of retinal vessels are initiated
  Other Names: Glyceryl Nitrate
Drug: COX-inhibitor + Nitroglycerin — Combination of COX-inhibitor and nitroglycerin interventions.

SUMMARY:
The primary objective is to study if a stimulation of nitric oxide and/or prostaglandin affect the diameter changes of retinal vessels during hypoxia. Diameter changes are studied using the Dynamic Vessel Analyzer.

ELIGIBILITY:
Inclusion Criteria:

* Age between >19 and <61 years
* No known systemic or ocular diseases

Exclusion Criteria:

* Cardio-vascular disease
* Lung disease
* Epilepsy
* Previous ocular disease
* Previous treatment with medications influencing the intraocular pressure or the metabolism of nitric oxide or prostaglandins
* Daily intake of medicine except contraceptive pills
* Pregnancy or breastfeeding
* Known allergy against any of the drugs used in the interventions

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-02; Primary Completion 2015-02 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Diameter changes of retinal vessels | Examination day 1 and 2
  Comparing the differences of diameter changes occuring during each of interventions

CONTACTS AND LOCATIONS:
Overall Officials: Line Pedersen, MD, Principal Investigator — Aarhus University Hospital; Musa Kaya, stud.med, Principal Investigator — Aarhus University Hospital
Locations (1):
- Department of Ophtalmology, Aarhus University Hospital, Aarhus, Denmark